CLINICAL TRIAL: NCT06247917
Title: A Prospective, Single-arm Clinical Study to Evaluate the Efficacy and Safety of Allogeneic Haematopoietic Stem Cell Transplantation With FLU-BU-MEL Conditioning for Myelodysplastic Syndromes
Brief Title: Evaluate the Efficacy and Safety of Allogeneic Haematopoietic Stem Cell Transplantation With FBM Conditioning for MDS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-2023-01
Record Dates: First submitted 2023-12-26; First posted 2024-02-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-12

CONDITIONS: Myelodysplastic Syndrome With Excess Blasts-1; Myelodysplastic Syndrome With Excess Blasts-2; Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — fludarabine; Busulfan; Melphalan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FBM group (Experimental): undergoing FBM regiment
  Interventions: Drug: Fludarabine, Busulfan and Melphalan

INTERVENTIONS:
Drug: Fludarabine, Busulfan and Melphalan — Use Fludarabine, Busulfan and Melphalan as myeloablative conditioning regimen for untreated MDS-EB patients.

SUMMARY:
To assess the safety and efficacy of FLU-BU-MEL as a conditioning regimen for allogeneic hematopoietic stem cell transplantation in patients with untreated MDS-EB or IPSS-R that is intermediate-risk (>3.5 points), high-risk, or very high-risk. The investigators conducted this clinical trial.There will be three phases to this trial: screening, therapy, and follow-up. A) Screening phase: Qualified patients are screened for trial participation by a medical history, physical examination, laboratory testing, and disease evaluation after providing their informed consent. B) Treatment duration: patients receive allogeneic hematopoietic stem cell transplantation prepped with Flu-Bu-Mel in accordance with the protocol. C) Follow-up period: patients were checked on at the scheduled time to assess safety and efficacy. HSCT conditioning regiment: Flu 30 mg/m2/d d-6 days to d-2 9 (intravenously over two hours), : MEL 50 mg/m2/d intravenously, d-3 to d-2; BU 0.8 mg/kg/q6h d-6 to d-5 (intravenously, over 2 hours per drip). Fludarabine and melphalan do not require a dose adjustment based on body weight; however, if body mass index BMI> 25, ideal body weight (IBW) should be calculated (as BMI=25), and then determine Busulfan dosage based on corrected body weight (AIBW25). AIBW25=IBW+25% x (actual body weight - IBW)

DETAILED DESCRIPTION:
The only curative treatment for myelodysplastic syndromes (MDS) is allogeneic hematopoietic stem cell transplantation (allo-HSCT), which is also the most likely means of extending survival in patients who are at higher risk. To maximize the survival advantage, it is uncertain whether higher-risk patients should receive allo-HSCT directly or whether it should be done after demethylation treatment or chemotherapy to lower the primitive cell count. According to retrospective investigations, patients did not experience an OS benefit with pre-transplantation demethylation therapy (Xixi Wang et al., China; G. Damaj et al., France)1，2. In contrast to sequential allo-HSCT with chemotherapy and demethylation, early allo-HSCT in patients with IPSS-scored high-risk/very high-risk MDS prolongs OS and improves survival, according to another meta-analysis3，4. There is currently only one available randomized trial that evaluated the two treatment regimens 5; however, it was prematurely stopped because of a delayed recruitment of patients 5. The Chinese recommendations for the Diagnosis and Treatment of Myelodysplastic Syndromes (2019 edition) and other international recommendations suggest that patients can have demethylation or chemotherapy without postponing transplantation, based on the evidence that is currently available. On the other hand, patients may be denied or delayed HSCT due to pre-transplant treatment toxicity.The traditional pretreatment strategy for myeloid tumors prior to transplantation was Busulfan with cyclophosphamide; however, in light of increased toxicity and treatment-related mortality, fludarabine (Flu)-based pretreatment regimens have increasingly taken the place of the former. Research indicates that patients treated with FluBu2/FluBu3 had a significantly lower percentage of T cells reaching complete donor chimerism within 30 days than patients treated with BUCY. Additionally, patients who achieve complete remission (CR) prior to transplantation have an overall survival (OS) rate of 50-80%, compared to 19-32% for those who do not achieve CR. Finally, the post-transplant recurrence rate can reach 50%.6, 7, indicating that FLU-BU is not recommended for individuals who are at high risk of recurrence and is not the best pretreatment regimen for immune reconstitution due to its limited antitumor impact. Thus, it is still a pressing problem to figure out how to boost the antitumor impact without making the pretreatment more hazardous.

Yamamoto et al reported the effectiveness of sequential single-copy cord blood transplantation for unremitting AML based on FLU-BU (FLU 30mg/m2/d*6d, BU 3.2mg/kg/d×4d) in combination with MEL 80mg/m2 as a pretreatment regimen 8, in order to investigate the possibility of obtaining a more optimal regimen. Out of 51 patients, 46 underwent implantation and attained full donor chimerism. The 2-year actual OS and progression-free survival (PFS) were 54.9%, the 2-year cumulative RI was 19.6%, the 100-day and 2-year cumulative NRM were 11.8% and 25.5%, respectively. indicating that there was no appreciable increase in toxicity and a greater antitumor efficacy with the MEL-enhanced FLU-BU regimen. For the purpose of treating AML/MDS, Tomoaki Ueda et al. introduced MEL 100 mg/m2 as a pretreatment regimen on top of FLUBU4 9. They demonstrated that all 42 patients were implanted and that full donor chimerism of T cells was attained in less than 30 days, 4 years: DFS 59.5%, NRM 19%, OS 66%. While the 5-year RI of 53.8% was present in 31% of these non-CR individuals, the group as a whole only had a 21.4% RI rate.In a multicenter, prospective research involving AML and MDS, Yoshimitsu Shimomura et al.10 evaluated allogeneic hematopoietic stem cell transplantation for hematological neoplasms pretreated with Flu/Bu4/Mel and Flu/Bu4 regimens. Propensity score was the primary factor that matched the two patient groups. The 5-year OS was higher in the Flu/Bu4/Mel group compared to the Flu/Bu4 group (32.4% vs. 30.1%, log-rank P = 0.019), and there was no significant difference between the two groups in terms of non-recurrent deaths. Additionally, the 5-year recurrence rate and recurrence-associated mortality rate were significantly lower in the Flu/Bu4 group than in the Flu/Bu4 group.

Based on prior research, the FLU-BU-MEL regimen appears to be workable for treating AML/MDS. It can also lower the rate of recurrence following allo-HSCT by providing a more potent anti-tumour effect and better implantation, while the treatment-related death rate is generally within an acceptable range and may even increase patient survival. In order to achieve this, a single-arm, open-ended, single-centre phase II clinical study is suggested. Its purpose is to assess the safety and effectiveness of the FLU-BU-MEL pretreatment regimen for the treatment of MDS in the untreated higher-risk group, as well as to serve as a foundation for a prospective future randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Myelodysplastic Syndromes (IB1/IB2)
2. Patients did not receive any anti-tumour therapy (including chemotherapy, immunotherapy (lenalidomide, etc.), targeted therapy, hormone therapy, etc.).

Exclusion Criteria:

1. CMML with 5q deletion or carrying PDGFRB fusion gene;
2. secondary MDS;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of relapse | 2 years
  2 years cumulative incidence of relapse

SECONDARY OUTCOMES:
Disease free survival | 2 years
  2 years Disease free survival
non relapse mortality | 100 days
  non relapse mortality within 100d of HSCT
non relapse mortality | 2 years
  non relapse mortality within 2 years of HSCT
cumulative incidence of acute graft-versus-host disease | 180 days
  180 days after HSCT
cumulative incidence of chronic graft-versus-host disease | 2 years
  2 years after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Luxiang Wang, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, China